CLINICAL TRIAL: NCT01156649
Title: Neurobehavioral Effects of Positive Airway Pressure (PAP) Therapy in Children With Obstructive Sleep Apnea
Brief Title: Effects of Positive Airway Pressure (PAP) in Children With Obstructive Sleep Apnea (OSA)
Acronym: OSA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-03572FB HL102151
Record Dates: First submitted 2010-07-01; First posted 2010-07-05 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; neurocognitive function; cognition; pediatrics; children; continuous positive airway pressure therapy; sham treatment; randomized clinical trial; behavior; treatment
MeSH Terms: conditions — Sleep Apnea, Obstructive; Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham PAP therapy (Sham Comparator): Sham PAP will be used with 30 children, and consists of continuous sub-therapeutic levels of air pressure (approximately 1 cm of water) that are delivered through the nasal interface device.
  Interventions: Device: Sham PAP therapy
- Treatment group (Active Comparator): 30 children will receive active treatment PAP, which consists of automatically adjusted air pressures that are delivered through the nasal interface device at levels which effectively treats the obstructive events.
  Interventions: Device: PAP therapy

INTERVENTIONS:
Device: PAP therapy — Nightly use of automatic positive airway pressure delivered at therapeutic levels and to be delivered through a nasal interface device selected to maximize comfort for each child.
  Other Names: CPAP; APAP; Continuous positive airway pressure therapy
  Arms: Treatment group
Device: Sham PAP therapy — During sleep, the sham PAP device will administer a constant pressure of subtherapeutic air (approximately 1 cm of water) through a custom fit nasal interface chosen for the child's maximum comfort.
  Other Names: CPAP; APAP; Continuous positive airway pressure therapy
  Arms: Sham PAP therapy

SUMMARY:
Obstructive sleep apnea is a problem for a large number of children and can result in problems with thinking patterns, behaviors and sleep if left untreated. Little is known about how positive airway pressure (PAP) therapy might help children who need treatment for obstructive sleep apnea. We will investigate how PAP therapy might be able to improve thinking patterns, behavior and sleep problems in children with obstructive sleep apnea.

DETAILED DESCRIPTION:
Positive airway pressure (PAP) therapy has been shown to be an effective treatment which can improve neurocognitive performance and sleep patterns in adults with obstructive sleep apnea (OSA). However, the effect of PAP therapy on neurocognitive, behavioral and sleep patterns in school-aged children with OSA is not well known. The goal of this innovative study is to conduct a randomized, double-blind, placebo controlled, trial which will determine the effects of PAP therapy on neurocognitive and behavioral patterns and sleep architecture in children with OSA. A battery of neurocognitive tests and parent behavioral rating assessments will be given to school-aged children with OSA before, after 3 months and again after 6 months of treatment with PAP therapy only; or 3 months of PAP placebo use followed by 3 months of PAP therapy. Full polysomnography and PAP titration sleep studies will be performed following a night of adaptation sleep in a sleep laboratory at all three time points. Compliance to PAP therapy will be monitored on a daily basis with a remote internet-linked communicator that is attached to the participant's PAP pressure generator. The hypothesis of this ground-breaking project is that 3 months of continuous compliance to a regimen of PAP therapy will result in significant improvement in neurocognitive and behavioral patterns and that sleep architecture will be positively changed to become more reflective of normative values for school-aged children. The results of this innovative and ground-breaking study will have far-reaching effects for sleep clinicians and other health care providers in support of the continued use of PAP therapy as a treatment for OSA and to inform the health-care community about the efficacy of PAP therapy on neurocognition and behavior patterns in school-aged children with OSA.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6.0 and 11.9 years
2. Nocturnal PSG (polysomnography) shows an apnea/hypopnea index of at least 1.5-10 events on average per hour of sleep and an apnea index of less than 1 per hour (mild to moderate OSA group), or, PSG shows an apnea index of 1 or greater PLUS an apnea/hypopnea index of 10.0 or greater (severe OSA group).
3. English is spoken as the child's primary language.
4. Willingness to complete study protocol if randomized into the placebo treatment group.

   -

Exclusion Criteria:

1. The presence of any other diagnosable sleep disorder other than OSA.
2. Previous use of PAP therapy for sleep disordered breathing at any time in the patient's history
3. Presence of health problems likely to interfere with neurocognitive test result interpretation, such as previously diagnosed psychiatric illness (i.e., attention-deficit hyperactivity disorder, depression, psychoses) or medical genetic syndromes (i.e., Prader-Willi syndrome, Fragile X).
4. Presence of a chronic neurological disorder, chronic renal failure, diabetes, rheumatoid arthritis, or another chronic inflammatory condition. -

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2010-07; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Neurobehavioral and cognitive function | 6-12 months
  a battery of tests designed to measure: academic achievement, reaction time, attention, working memory, executive function, decision making and mental flexibility, and fine motor speed and coordination.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen H Archbold, PhD, RN, Principal Investigator — University of Tennessee Health Science Center College of Nursing
Locations (1):
- LeBonheur Pediatric and Adolescent Sleep Disorders Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No